CLINICAL TRIAL: NCT00359398
Title: Post-operative Administration of Platelet Rich Plasma Sequestered Prior to Cardiopulmonary Bypass Reduces the Coagulopathy Associated With Complex Cardiac Surgery
Brief Title: Sequestration of Platelets Prior to Bypass Reduces Bleeding After Cardiac Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding expired, low recruitment
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006IC003B
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Cardiac Surgical Procedures; Cardiopulmonary Bypass; Blood Platelet Disorders; Blood Coagulation Disorders
Keywords: Cardiopulmonary bypass; Blood component removal
MeSH Terms: conditions — Blood Platelet Disorders; Blood Coagulation Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet sequestration (Experimental): Sequestration of platelet rich plasma before cardiopulmonary bypass
  Interventions: Procedure: Platelet rich plasma sequestration
- Standard care (No Intervention): No platelet rich plasma sequestration undertaken before cardiopulmonary bypass (usual practice)

INTERVENTIONS:
Procedure: Platelet rich plasma sequestration — Venesection of blood (14 ml/kg) and separation to red cells and platelet rich plasma.
  Other Names: Haemonetics cell salavage system
  Arms: Platelet sequestration

SUMMARY:
Excessive bleeding is common after cardiac surgery. This may result in patients receiving a blood transfusion or suffering the life-threatening complication of cardiac tamponade. Tamponade is when excessive bleeding compresses the heart and prevents it from pumping properly. A major reason for the bleeding is the damage done to platelets by the cardiopulmonary bypass (CPB) machine. Often patients receive platelets and plasma from blood donors to try to reduce the bleeding post-operatively. The investigators plan to take platelets and plasma from patients before they are damaged. They would then return these 'undamaged' sequestered platelets to the patients after the bypass machine is no longer needed. Therefore, the investigators' primary question is whether platelet sequestration would reduce the bleeding problems that occur following cardiac surgery. They will evaluate bleeding problems using thromboelastography, which provides a comprehensive assessment of both how blood clots form and their strength. If sequestration reduces bleeding problems following cardiac surgery then it may reduce the chance of patients receiving blood products from donors. Although donated blood is thoroughly tested, its use does expose patients to the risk of transfusion errors, blood borne infections and reactions. Avoiding its use would be very desirable.

DETAILED DESCRIPTION:
Hypothesis:

Patients undergoing repeat median sternotomy or requiring prolonged cardiopulmonary bypass (CPB) often develop a coagulopathy at the end of surgery. We propose sequestering plasma and platelets from these patients prior to CPB and thus prior to the dilution and platelet damage that occurs with CPB. We hypothesise that if these plasma and platelets are stored properly during CPB, and administered at the end of the operation, they will reduce any coagulopathy and the associated bleeding.

Study population:

Patients undergoing repeat median sternotomy, mitral valve repair, double valve operations, aortic surgery, or combined valve and coronary artery surgery.

Exclusion criteria will include those with anaemia, thrombocytopenia, unstable angina, anti-platelet therapy within the previous seven days, known or symptomatic cerebrovascular disease, known disorders of haemostasis, aprotinin sensitivity and pregnancy.

Intervention:

Patients will be randomised by a closed envelope technique to receive platelet/plasma sequestration or not. Patients randomised to undergo sequestration will have 14 mL/Kg blood taken. The blood will be separated into red cells and platelets/plasma. Anaemia would be prevented by returning the processed red blood cells to the patient. We will store platelets at 20-24°C/room temperature on a platelet rocker according to guidelines from the National Blood Service.

Assessment of coagulation:

Patients' coagulation status will be evaluated before and after surgery. Four methods will be employed to comprehensively assess the coagulation system: platelet counts and conventional clotting studies; heparin levels; thromboelastography; and platelet function analyser.

ELIGIBILITY:
Inclusion Criteria:

Adult patients undergoing cardiac surgery that involves:

* Repeat median sternotomy
* Mitral valve repair
* Double valve operations
* Combined valve and coronary surgery
* Anticipated prolonged cardiopulmonary bypass

Exclusion Criteria:

* Pre-operative anaemia
* Pre-operative thrombocytopenia
* Unstable angina
* Anti-platelet therapy (e.g. aspirin, clopidogrel) within the previous 7 days
* Known or symptomatic cerebrovascular disease
* Known disorders of haemostasis
* Aprotinin sensitivity
* Pregnancy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Incidence of coagulation abnormalities as assessed by thromboelastography and platelet function analyser | At end of surgery (usually <1 day)

SECONDARY OUTCOMES:
Volume of blood lost into chest drains during first 24 post-operative hours | 24 hours
Volume of blood product administered during first 24 post-operative hours | 24 hours
Length of stay in the intensive care unit (ICU) | Usually < 30 days
ICU mortality | Usually < 30 days
Incidence of surgical re-exploration | Hospital admission (usually < 30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Simon J Finney, MBChB, PhD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust; Andrea Kelleher, MBBS, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust; Judith Hall, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust; Simon Davidson, PhD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom